CLINICAL TRIAL: NCT03486249
Title: Interaction Between Diaphragm and Cardiac Function During Weaning From Mechanical Ventilation
Brief Title: Interaction Diaphragm and Cardiac Function During Ventilator Weaning
Acronym: I-DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K180103J
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Ventilator Weaning
Keywords: diaphragm dysfunction; ventilator weaning; pulmonary edema
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Intervention Model Description: All patients will have a cardiac echo examination and diaphragm function assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient difficult to wean (Experimental): Repetition of medical examinations performed as part of the care. All patients will have a cardiac echo examination and diaphragm function assessment before the spontaneous breathing trial.
  Interventions: Other: Repetition of medical examinations performed as part of the care

INTERVENTIONS:
Other: Repetition of medical examinations performed as part of the care — Cardiac echo, diaphragm ultrasound and phrenic nerves stimulation performed before the spontaneous breathing trial.

SUMMARY:
Weaning failure is associated with prolonged duration of mechanical ventilation that itself can worsen patient's prognosis. Therefore, identification of the causes and mechanisms leading to weaning failure is important in daily practice. While diaphragm dysfunction and pulmonary edema are two main causes of weaning failure, there are currently no data that quantify their respective contribution neither their potential co-existence. During weaning from mechanical ventilation, heart and lung interaction plays a major role. As a key factor, diaphragm function is therefore certainly involved in the occurrence of weaning-induced pulmonary edema. However, both phenomenons diaphragm dysfunction and weaning induced pulmonary edema have not been simultaneously investigated so far. This current project aims at exploring the relationship between diaphragm dysfunction and pulmonary in patients experiencing weaning failure. The objectives are 1) to quantify the respective contribution and co-existence of diaphragm dysfunction and weaning induced pulmonary edema and 2) to investigate the role of diaphragm function in the occurrence of weaning induced pulmonary edema.

DETAILED DESCRIPTION:
The study will take place in the Medical ICU of Pitié-Salpêtrière Hospital in Paris. The ICU have an established and successful clinical research program and infrastructure.

ICU patients will be enrolled if eligible (based on inclusion and non inclusion criteria) after their first spontaneous breathing trial failure.

Diaphragm function will be assessed by its capacity to generate a pressure with the phrenic nerves stimulation technique (reference method) and by ultrasonography (thickening fraction). Weaning induced pulmonary edema will be diagnosed with cardiac echo and markers of plasma contraction (plasma protein concentration).

Phrenic nerves stimulation, diaphragm and cardiac ultrasound will be repeated as part of the research before the spontaneous breathing trial.

After obtaining consent and before starting the second spontaneous breathing trial, clinical and biological will be collected. EKG and maximal inspiratory pressure will be done. Then, a diaphragm ultrasound and cardiac echo will be done and the phrenic nerves stimulation method will be undertaken. After these measurements, the spontaneous breathing trial will start. At the end of the spontaneous breathing trial (30 minutes with pressure support 7 cmH2O and 0 positive end expiratory pressure) or sooner in case of intolerance (respiratory distress), a new cardiac echo and diaphragm ultrasound will be performed as part of standard care before resuming the initial ventilator settings. As recommended by the usual medical practice, a second phrenic nerves stimulation will be eventually done after resuming the initial ventilator settings.

Diaphragm capacity to generate pressure :

Twitch airway pressure (Ptr, stim) will be measured during phrenic nerve stimulation. Phrenic nerve stimulation will be performed by bilateral anterior magnetic stimulation.

Cardiac echo :

Cardiac echo will be performed with a Philips Sparq ultrasound with a dedicated probe. The following variables will be obtained: left ventricular ejection fraction, E wave, A wave, E' wave, TAPSE

Diaphragm ultrasound :

Diaphragm thickening fraction will be measured by placing 13 MHz transducer on the right chest wall in the ninth intercostal space mid-way between the anterior and mid-axillary line and held perpendicular to the chest wall. Thickening fraction will be computed as the percentage change in thickness between end-expiration (i.e. minimum muscle thickness) and peak inspiration (i.e. maximal muscle thickness) visualized in M-mode.

ELIGIBILITY:
Inclusion Criteria:

1. Patients adult (age ≥ 18 years)
2. Intubation and invasive mechanical ventilation longer than 48 hours;
3. Failure to the first spontaneous breathing trial;
4. Presence of weaning readiness criteria
5. Oral informed consent
6. Patient with affiliation to the french healthcare system

Exclusion Criteria:

1. Pregnant women
2. Patient opposition
3. Contraindication to perform magnetic phrenic nerves stimulation technique (chest tube, cardiac pacemaker or implanted defibrillator, cervical implants, chest drains,...)
4. Impossibility to consider ventilator weaning (total ventilator dependence : preexisting neuromuscular disorders, cervical spine injury…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Failure at the spontaneous breathing trial | During or at the end of the spontaneous breathing trial
  Weaning failure defined by the criteria of the International Conference on Weaning (Boles et al. ERJ 2007)

SECONDARY OUTCOMES:
Rate of patients with diaphragm dysfunction | At the end of the patient participation (Day 3)
  Diaphragm dysfunction will be defined as a decrease capacity of the diaphragm to generate a pressure
Rate of patients with weaning induced pulmonary edema | At the end of the patient participation (Day 3)
  Weaning induced pulmonary edema will be defined by an increase in left filling pressure and/or plasma protides concentration
Rate of patients with diaphragm dysfunction and weaning induced pulmonary edema | At the end of the patient participation (Day 3)
  Diaphragm dysfunction will be defined as a decrease capacity of the diaphragm to generate a pressure and weaning induced pulmonary edema will be defined by an increase in left filling pressure and/or plasma protides concentration

CONTACTS AND LOCATIONS:
Overall Officials: Martin DRES, MD, PhD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Paris, France